CLINICAL TRIAL: NCT04059263
Title: Impact of Hexafluoroisopropanol (HFIP) on the Inflammatory Response in Blood of Septic Patients (HFIP Ex-vivo Study). A Feasibility, Proof of Principle Project.
Brief Title: HFIP Ex-vivo Study
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2019 - 00774
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sepsis, a multi organ failure caused by infectious diseases, is a major health burden with an average mortality rate of 26%. Cells of the innate immune system of hosts recognize specific patterns of pathogenic bacteria and trigger an inflammatory response. In case of sepsis, this inflammatory response takes a deregulated course, expressing an overwhelming amount of pro-inflammatory cytokines leading to a loosening of endothelial tight junctions, evasion of intravasal fluids and proteins into the interstitium, as well as direct tissue damage throughout an overproduction of reactive oxygen species by neutrophils. These pathological changes of the host's proper immune system lead to a multi organ failure, which characterize a clinical pathomechanism of sepsis. Several studies confirmed an immunomodulatory effect of sevoflurane's primary metabolite hexafluoroisopropanol (HFIP) attenuating pro-inflammatory cytokine expression with a consecutive improvement of organ function and survival in rodent models of sepsis. Until now, there are no data available confirming this effect in septic patients as well. With this study, the direct impact of sevoflurane's primary metabolite HFIP on cytokine expression in the blood of septic patients will be investigated for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency ward with suspicion of infection and a qSOFA Score ≥ 2 points (Respiratory frequency > 22/minute, Systolic blood pressure < 100 mmHg, Glasgow Coma Scale < 15).
* Male and Female subjects with at least 18 years of age.
* Written informed consent by the participant after information about the project. In emergency cases where a written consent cannot be obtained immediately, due to the patient's medical conditions, the existence of a patient decree and of a representative in the emergency situation is evaluated according to the Swiss Civil Code. Informed consent will be obtained from the representative. A medical doctor, furthermore, not participating in the investigation, guarantees the medical care of the patient by the defending of his/her interests. After recovery, the patient will be informed as soon as possible about the trial and consent is requested.

Exclusion Criteria:

* Acquired Immune Deficiency Syndrome
* Anti-IL-6 therapy (e.g. Kevzara®) within the last 60 days
* Application of a cytokine absorber
* Pregnancy and/or Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the emergency department of tertiary care hospital with suspicion of an infection and a qSOFA score ≥ 2 points.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Inflammatory response in blood of septic patients after application of HFIP | IL-6 will be measured after 6 hours incubation.
  Interleukine-6 (IL-6) will be measured with Enzyme-linked Immunosorbent Sandwich Assay as a surrogate marker of inflammatory response. Amount of IL-6 is compared between treated samples and control samples.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Beck Schimmer, Prof. Dr. med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No